CLINICAL TRIAL: NCT00638469
Title: Prospective, Randomized Half-side Study on the Efficacy of UVB-311nm Phototherapy in Patients With Psoriasis After Partial Remission to Treatment With Adalimumab
Brief Title: UVB-311nm After Initial Slow Response to Adalimumab in Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Professor of Bioimmunotherapy, Medical University of Graz
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-133 ex 07/08
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Psoriasis
Keywords: Psoriasis; Biologic; adalimumab; narrowband UVB; phototherapy; half-side comparison
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- left/right (Other): left or right body side
  Interventions: Radiation: UVB-311nm; Other: No treatment

INTERVENTIONS:
Radiation: UVB-311nm — UVB-311nm radiation given 3 times a week to one randomized body half
  Other Names: narrow-band UVB radiation
Other: No treatment — no UV exposure

SUMMARY:
Adalimumab, a fully human anti-tumor necrosis factor (TNF) monoclonal antibody has been approved for the treatment of moderate to severe psoriasis. However, in a portion of cases adalimumab does not induce reduction of psoriasis area and severity index (PASI) of 75% or greater, now being considered as gold standard for treatment efficacy. In this study we aim to determine in a randomized half-side comparison whether additional narrowband UVB-311nm phototherapy accelerates and improves the clearance of psoriatic lesions in adalimumab-treated patients after initial slow response.

DETAILED DESCRIPTION:
Patients with moderate to severe psoriasis who have received treatment with adalimumab (loading dose of 80 mg and thereafter 40 mg s.c. biweekly) for at least 6 weeks without a PASI reduction of 75% or greater qualify for the study. Adalimumab is continued and UVB-311nm phototherapy is added at 6 weeks or thereafter one a randomized body half (left or right; head exempt) 3 x per week until complete response (defined as reduction in PASI to < 3) for a maximum of another 6 weeks (until week 12). PASI score, visual analogue score (VAS) patient score for therapeutic response, and VAS patient score for severity of skin lesions is assessed weekly; and at follow-up visits at month 3, 6, and 12. Paired Wilcoxon testing for differences in PASI and patient VAS scores is done; Fischer exact test is applied to determine differences in complete remission, PASI reduction > 90%, > 75% and/or 50% between body sites.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis patients with PASI reduction of less than 75% after at least 6 weeks of treatment with adalimumab.

Exclusion Criteria:

* Pregnancy or lactation
* History of skin cancer
* Presence of or history of malignant skin tumors
* Dysplastic melanocytic nevus syndrome
* Antinuclear antibodies (ds-DNA, Ro/SSA, La/SSB)
* Autoimmune disorders such as Lupus erythematosus or Dermatomyositis
* Photosensitive diseases such as porphyria, chronic actinic dermatitis, Xeroderma pigmentosum, basal cell nevus syndrome, and others
* General poor health status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Modified PASI (psoriasis area and severity index) | 12 months

SECONDARY OUTCOMES:
VAS patient score for therapeutic effect | 12 months
VAS patient score for severity of skin lesions | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Medical University of Graz, Department of Dermatology, Graz, Austria